CLINICAL TRIAL: NCT05069662
Title: Assessment of the Impact of the COVID-19 Pandemic on Drug Use and on the Perception of Remote Monitoring by Cancer Patients Followed in the ONCORAL Program
Brief Title: Impact of the COVID-19 Pandemic on Drug Use and Monitoring of Cancer Patients
Acronym: ONCORAL-Covid
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0163
Record Dates: First submitted 2021-10-04; First posted 2021-10-06 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cancer
Keywords: remote monitoring; oral anticancer drugs; drug intake; COVID-19 pandemic
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with oral anticancer drugs: Patients treated with oral anticancer drugs followed in the Oncoral program
  Interventions: Other: Directive Interview

INTERVENTIONS:
Other: Directive Interview — One directive interview conducted by telephone

SUMMARY:
The COVID-19 pandemic has profoundly changed the organisation of care. Teleconsultation has replaced hospital medical consultations in order to reduce the risk of patient exposure to the virus.

Within the framework of the Oncoral multidisciplinary outpatient / hospital program of follow-up, carried out by the Hospices Civils de Lyon for ambulatory patients treated with oral anticancer drugs, interviews with the pharmacist and/or nurse, which were previously organised face-to-face, have been replaced by telephone interviews, ensuring continuity of follow-up for patients without having to come to the hospital.

This study focuses on a telephone survey to describe the impact of the COVID-19 pandemic health crisis on the drug exposure of cancer patients followed in the Oncoral program, their treatment management, their perception of teleconsultation and their IT resources for remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 and over
* Ambulatory patients treated with oral anticancer drugs and benefiting from the ONCORAL multidisciplinary outpatient / hospital program
* Having benefited from a remote monitoring between March 16, 2020 and May 11, 2020 (the COVID-19 pandemic-related containment period)
* Patients who do not object to participating in the survey and to the use of the data collected

Exclusion Criteria:

* Patients who do not speak French
* Patients living in an institution
* Patients protected by law
* Patients included in a drug clinical trial
* Patients refusing to participate in the survey and / or not responding to the 2 telephone calls requesting their participation and / or not responding to any of these calls
* Patients choosing to stop the interview and no longer answering to the questions asked

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with oral cancer drugs included in the Oncoral multidisciplinary outpatient / hospital program of the Hospices Civils de Lyon and having benefited from remote monitoring during the COVID-19 pandemic-related containment period between March 16, 2020 and May 11, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reporting a change in drug use during the COVID-19 pandemic-related containment period. | Inclusion
  Percentage of patients reporting a change in medication use and / or a change medication management and / or a change in oral anticancer drug adherence during the COVID-19 pandemic-related containment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Service Pharmaceutique, Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No